CLINICAL TRIAL: NCT06853951
Title: The Effect of Cardioprotective Medications on Chemotherapy-Induced Cardiotoxicity in Childhood Acute Leukemia
Brief Title: Cardioprotection on Chemotherapy-Induced Cardiotoxicity
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, keristin nazir, Teaching Assistant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 315
Record Dates: First submitted 2025-02-21; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Cardiotoxicity
MeSH Terms: conditions — Cardiotoxicity | interventions — Angiotensin-Converting Enzyme Inhibitors; Captopril; Carvedilol

STUDY DESIGN:
Intervention Model Description: Arm 1 Patients will receive ACEIs oral tablets during Induction Phase by either a caregiver or caring nurse.
  Arm 2 Patients will receive β-blockers oral tablets during Induction Phase by either a caregiver or caring nurse.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACEIs (Active Comparator): 0.3 mg/kg/dose every 8 hours orally by either a caregiver or caring nurse.
  Interventions: Drug: ACE Inhibitors
- β-blockers (Active Comparator): 0.05 mg/kg/dose every 12 hours orally by either a caregiver or caring nurse
  Interventions: Drug: β -Blockers

INTERVENTIONS:
Drug: ACE Inhibitors — 0.3 mg/kg/dose every 8 hours orally by either a caregiver or caring nurse.
  Other Names: Captopril
  Arms: ACEIs
Drug: β -Blockers — 0.05 mg/kg/dose every 12 hours orally by either a caregiver or caring nurse.
  Other Names: Carvedilol
  Arms: β-blockers

SUMMARY:
The aim of the present study is to evaluate the protective impact of cardioprotective medications on the chemotherapy- induced cardiotoxicity.

DETAILED DESCRIPTION:
The goal of this interventional study is to evaluate the protective impact of Angiotensin-converting enzyme (ACE) inhibitors versus β-blockers on the cardiotoxicity profile of pediatric patients with acute leukemia. The impact is measured by evaluation of left ventricular ejection fraction (LVEF) by 2D echocardiography at baseline and at the end of Induction phase (42 days).

ELIGIBILITY:
Inclusion Criteria:

* Willingness of the legal representative of research participant to participate in the study by giving "informed consent."
* Ability to take oral medication.
* Age 2-18 years at the time of diagnosis.

Exclusion Criteria:

* Documented allergy to cardioprotective medications

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-07-18 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (LVEF) | LVEF will be measured at Baseline and at the end of Induction Phase (42 Days)
  he LVEF will be measure by 2D Echocardiography at baseline and at the end of Induction Phase (42 Days)

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hamed El-Hamamsy, Prof, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Pharmacy, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes